CLINICAL TRIAL: NCT02525250
Title: Pilot Study Immunomonitoring NK Cells in Patients With Myeloid Malignancies
Brief Title: Pilot Study Immunomonitoring Natural Killers Cells in Patients With Myeloid Malignancies Treated With Lenalidomide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MDS-AML-NK / IPC-2012-007
Record Dates: First submitted 2013-04-03; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Acute Myeloid Leukemia or Myelodysplasic Syndrome
Keywords: Acute myeloid leukemia or myelodysplasic syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute myeloïd leukemia (Experimental): Realization of 3 blood samples at day 0, day 15 and day 28.
  Interventions: Procedure: Realization of 3 Blood samples during study during treatment with lenalidomide

INTERVENTIONS:
Procedure: Realization of 3 Blood samples during study during treatment with lenalidomide

SUMMARY:
This project is a framework for developing new therapeutic strategies for acute myeloid leukemia(AML)based immunotherapy.

the role of NK cells was demonstrated in AML and especially GVL effect (graft versus leukemia) during allogeneic transplantation in these patients. However, it has been shown that the phenotype of NK cells and their cytotoxic functions were altered during this malignancy. In addition, in these patients, impaired NK function is associated with relapse.

lenalidomide it would have a beneficial effect on NK cells of AML patients? Does it have a role in leukemic cells in this malignancy? what is its effect on the production of pro-inflammatory cytokines? In vitro data show an effect of lenalidomide on the phenotype of NK cells from healthy donors and patients with LAM, and despite these phenotypic changes, the cytotoxic capacity of NK is not altered.Lenalidomide also induces a significant increase in the production of TNF-alpha (tumor necrosis factor) by NK.

It also seems to have an effect on leukemic blasts of AML. So, the investigators hope this study confirm these results in vivo in peripheral blood cells in patients treated with lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and above,
* Patient with myeloid acute leukemia or with myelodysplasic syndrome, treated or should be treated with Revlimid,
* Signed consent to participate,
* Patient affiliated to a social security system or benefiting from such as a system.

Exclusion Criteria:

* Allogeneic patients beyond,
* Patient deprived of liberty or under supervision of a guardian,
* Impossibility to undergo medical examinations of the study for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of NK functions | Time from inclusion (Day 0) until Day 28
  Evaluation with blood analysis

SECONDARY OUTCOMES:
cytotoxic response therapy | Time from inclusion until relapse or death (until 5 years)
  Evaluation of cytotoxic response therapy with lenalidomide

CONTACTS AND LOCATIONS:
Overall Officials: Thomas PREBET, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Thomas PREBET, MD, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr